CLINICAL TRIAL: NCT01560130
Title: Using a State-wide Initiative to Disseminate Effective Behavioral Weight Loss Strategies
Brief Title: State-wide Health Approach to Increase Reach and Effectiveness: Study 2
Acronym: SHARE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Rena R. Wing, Professor, The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 211699-7; R18DK083248 (NIH)
Record Dates: First submitted 2012-03-20; First posted 2012-03-22 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Population Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Shape Up Rhode Island + Online Weight Loss + Incentives (Active Comparator)
  Interventions: Behavioral: Shape Up Rhode Island + Online weight loss + Incentives
- Shape Up Rhode Island + Online weight loss program (Active Comparator)
  Interventions: Behavioral: Shape Up Rhode Island + Online weight loss program
- Shape Up Rhode Island + Online weight loss program + groups (Active Comparator)
  Interventions: Behavioral: Shape Up Rhode Island + Online weight loss program + Groups

INTERVENTIONS:
Behavioral: Shape Up Rhode Island + Online weight loss program — Participants assigned to this arm will receive the standard Shape Up Rhode Island statewide intervention and an Internet-based behavioral weight loss program.
  Arms: Shape Up Rhode Island + Online weight loss program
Behavioral: Shape Up Rhode Island + Online weight loss program + Groups — Participants assigned to this arm will receive the standard Shape Up Rhode Island statewide intervention, an Internet-based behavioral weight loss program, and the option to attend group sessions.
  Arms: Shape Up Rhode Island + Online weight loss program + groups
Behavioral: Shape Up Rhode Island + Online weight loss + Incentives — Participants assigned to this arm will receive the standard Shape Up Rhode Island statewide intervention, an Internet-based behavioral weight loss program, and monetary incentives for submitting self-monitoring information and for achieving clinically significant weight loss.
  Arms: Shape Up Rhode Island + Online Weight Loss + Incentives

SUMMARY:
Behavioral weight loss programs can successfully reduce body weight, but these programs are available to limited numbers of overweight and obese individuals. This project evaluates a unique weight loss approach that combines a self-sustaining weight loss campaign (for outreach) with training in behavioral weight loss strategies and tests the efficacy of adding components designed to enhance accountability and increase motivation for weight loss.

DETAILED DESCRIPTION:
This is a randomized trial. Participants will be randomly assigned to 1 of 3 treatment arms: (1) Shape Up Rhode Island (a community-based weight loss campaign) plus and Internet-based behavioral weight loss program (SURI+IBWL), (2) SURI + IBWL + optional group sessions (SURI+IBWL+Group), or (3) SURI+IBWL + monetary incentives for submitting self-monitoring information and achieving clinically significant weight loss. The primary outcome is weight loss at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index >=25 kg/m2
2. English speaking

Exclusion Criteria:

1. Health problems that make weight loss or unsupervised exercise unsafe
2. Current pregnancy or plan to become pregnant in the next 12 months
3. Planned relocation
4. Previous participation in Shape Up Rhode Island research studies

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2012-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Weight change from the initial assessment to the 3-month follow-up assessment measured on a digital scale to the nearest 0.1-kilogram | 0 to 3 months

SECONDARY OUTCOMES:
Weight change from the initial assessment to the 6-month assessment measured on a digital scale to the nearest 0.1-kilogram | 0 to 6 months
Weight change from the initial assessment to the 12-month assessment measured on a digital scale to the nearest 0.1-kilogram | 0 to 12-months

CONTACTS AND LOCATIONS:
Overall Officials: Rena R Wing, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- The Miriam Hospital's Weight Control and Diabetes Research Center, Providence, Rhode Island, United States